CLINICAL TRIAL: NCT02636816
Title: Cardiovascular Effects of Carbetocin During Elective Caesarean Delivery: A Randomized Controlled Trial Comparing Infusion Versus Bolus Administration Using Nexfin™
Brief Title: Cardiovascular Effects of Carbetocin Given During Elective Cesarean
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: H15-03007
Record Dates: First submitted 2015-11-30; First posted 2015-12-22 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Effect of Carbetocin on Cardiovascular System; Pregnancy
MeSH Terms: interventions — carbetocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infusion (Experimental): carbetocin is given slowly
  Interventions: Drug: carbetocin
- Bolus (Active Comparator): carbetocin is given quickly
  Interventions: Drug: carbetocin

INTERVENTIONS:
Drug: carbetocin — drug used to increase the tone of uterine muscle to prevent post partum hemorrhage after cesarean delivery.
  Other Names: Duratocin

SUMMARY:
The investigators are investigating whether slow administration of carbetocin is tolerated by patients better than if it is administered quickly, with respect to side effects such as headache, nausea, vomiting and facial flushing.

DETAILED DESCRIPTION:
Patients undergoing elective cesarean under spinal are included in the study. These patients are treated with carbetocin to reduce blood loss from the lining of the womb after delivery of the baby. The study is a randomised double blind controlled trial with 2 groups. One group will receive carbetocin quickly, the second group will receive carbetocin slowly. The investigators will compare the difference between groups with respect to side effects and the effect of carbetocin on the cardiovascular system.

ELIGIBILITY:
Inclusion Criteria:

* elective cesarean delivery under spinal,
* low risk for post partum hemorrhage,
* able to understand english

Exclusion Criteria:

* cesarean under general anesthesia,
* bleeding condition,
* placenta previa,
* unable to understand english

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
percent change in cardiac output parameters as measured by non-invasive cardiac output monitor | 10 minutes
  the parameters will be presented as percentage change from the baseline, which is determined prior to the start of the study period

SECONDARY OUTCOMES:
incidence of side effects occurring within timeframe below | 30 minutes
  headache, nausea, vomiting, facial flushing

CONTACTS AND LOCATIONS:
Overall Officials: Vit Gunka, MD FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada